CLINICAL TRIAL: NCT06603337
Title: Sequencing in Inflammatory Bowel Diseases (IBD) Therapy: "the Latium Net". A Key Multicenter Study
Brief Title: Sequencing in Inflammatory Bowel Diseases (IBD) Therapy: "the Latium Net".
Acronym: STRIKE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: STRIKE - 6837
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: IBD (Inflammatory Bowel Disease)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients treated with IBD from January 2015 to June 2024 will be included
- Prospective cohort: Consecutive patients with IBD who are starting, from clinical practice, new biologic/small molecule therapies, "failure" (already exposed) to a mechanism of action (for anti TNF-alpha, multiple molecules are allowed), and who belong to the Lazio Regional Health System will be enrolled.

SUMMARY:
Patients with IBD, both UC and CD, who fulfil the inclusion and exclusion criteria will be included consecutively:

* Retrospective cohort Patients treated with IBD from January 2015 to June 2024 will be included.
* Prospective cohort Consecutive patients with IBD who are starting, from clinical practice, new biological/small molecule therapies, failure (already exposed) to a mechanism of action (for anti TNF-alpha, more than one molecule is allowed), and who belong to the Lazio Regional Health System.

Eligible subjects will be identified among patients belonging to the IBD Unit of the Digestive Diseases Centre (CEMAD) of the Foundation and to all the other IBD Units of all the centres specified in Annex 1. Based on the number of patients referred to the clinics, we estimate 112 patients per month, the time for recruitment is 24 months.

Potential study participants will receive oral and written information about the study. Patients who agree to participate in the study will be asked to sign a written informed consent according to GCP.

DETAILED DESCRIPTION:
Multicenter, ambispectic observational study with drug

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years
2. Patients with a previous diagnosis of CD or UC at least 3 months before baseline.
3. Patients who have already failed at least one advanced (biological or small molecule) therapy for IBD and who have experienced failure to at least one mechanism of action (failure is defined as primary failure, secondary failure, or intolerance).
4. Patients who have already started a new advanced therapy for IBD based on clinical practice indication (primary loss of response, secondary loss of response, intolerance to the previous drug) since at least 1 week and up to 8 weeks after starting it.
5. Written informed consent certifying the willingness of the subject to participate to the study.

Exclusion Criteria:

1. Age < 18 years.
2. Patients with diagnosis of indeterminate colitis.
3. Patients naive to advanced (biological or small molecule) therapy for IBD.
4. Refusal to sign written informed consent certifying the willingness of the subject to participate to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IBD, both UC and CD, who meet the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Steroid-free deep remission of IBD | 24 months
  To evaluate the percentage of patients achieving the steroid-free deep remission of UC and CD after 12 months of different II line therapy (second sequential biological/advanced therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Franco Scaldaferri, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC CEMAD, Roma, Italy

IPD SHARING:
Plan to Share IPD: No